CLINICAL TRIAL: NCT01776866
Title: Comparison of Image Content Assessment Between Dural-axis Rotational and Standard Coronary Angiography
Brief Title: Image Content Analysis of Dural-axis Rotational Versus Standard Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20130101; 20130101 (Other: General hospital of CAPF)
Record Dates: First submitted 2013-01-16; First posted 2013-01-28 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Angiography; Rotational Coronary Angiography; Contrast Media; Radiation; Quantitative Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Coronary Angiography (Other): Patient first undergo standard coronary angiography(SA) of either left or right coronary system followed by dual-axis rotational coronary angiography(DARCA). The SA protocol consist of six different projections (right anterior oblique (RAO)-caudal, RAO-cranial (CRA), left anterior oblique (LAO)-CRA, LAO-caudal (CAU), antero-posterior (AP)-CRA and AP-CAU) for left coronary artery (LCA) and two projections (LAO and AP-cranial) for right coronary artery (RCA).
  The DARCA protocol consist of two coronary acquisitions specified by the protocol: one for LCA (Swing LCA CRA 35 5.8s), another for RCA (Swing RCA AP 4.0s).
  Interventions: Procedure: Coronary Angiography

INTERVENTIONS:
Procedure: Coronary Angiography — Coronary angiography include standard coronary angiography (SA) and dual-axis rotational coronary angiography (DARCA). Patient first undergo SA of either left or right coronary system followed by DARCA.

SUMMARY:
The investigators hypothesized that dual-axis rotational coronary angiography was non-inferior to standard coronary angiography with respect to diagnosis of coronary artery disease.

DETAILED DESCRIPTION:
The prior studies have demonstrated that dual-axis rotational coronary angiography (DARCA) is associated with lower contrast usage and radiation exposure compared with standard coronary angiography (SA). Single-axis rotational coronary angiography (RA) has been proved by previous studies without any reduction in diagnostic accuracy compared to SA. However, the rotational protocol is obvious different between DARCA and single-axis RA. A recent study has assessed the diagnostic accuracy of DARCA, but this study was not designed for image content analysis and the number of patients included did not provide sufficient statistical power to allow a valid comparison of DARCA with SA. The diagnostic accuracy of DARCA aroused our attention.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old, <80 years old
* a clinical indication for diagnostic coronary angiography to evaluate possible coronary artery disease

Exclusion Criteria:

* Pregnancy
* Known allergy to iodinated contrast
* Patients who had received iodinated contrast material within the last week or were unable to give consent
* Renal insufficiency (>1.5mg/dL)
* Acute myocardial infarction within one week
* Cardiogenic shock
* heart function worse than New York Heart Association functional class III
* Left main coronary artery disease
* Prior coronary artery bypass graft treatment
* Prior percutaneous coronary intervention treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Coronary Heart Disease | After coronary angiography, an expected average of 1 month
  The number of patients diagnosed as coronary heart disease by either angiographic modality by two blinded independent reviewers are recorded. The single criterion for diagnosis of coronary heart disease is the presence of coronary artery stenoses greater than or equal to 50%.

SECONDARY OUTCOMES:
Coronary Lesion Assessment | After coronary angiography, an expected average of 1 month
  The number of lesions greater than or equal to 50% detected by either angiographic modality by two blinded independent reviewers are recorded. In addition, they are asked to comment on the characteristics of the greater than or equal to 50% lesions (number of coronary lesions, number of bifurcation lesions, location of lesion, multivessel disease, American College of Cardiology (ACC) lesion classification and Medina classification for bifurcation lesions)
Quantitative Coronary Angiography | After coronary angiography, an expected average of 1 month
  The quantitative coronary angiography analysis of the more than or equal to 50% lesions detected by the lesion assessment of either reviewer one or reviewer two in both angiographic modalities (lesion length, minimum lumen diameter, diameter stenosis). Quantitative coronary angiography analysis will be performed by the third different blinded, independent, reviewer.
Diagnostic Screening Adequacy | After coronary angiography, an expected average of 1 month
  Two different experienced reviewers analyzed the angiographic sets based on a Likert Scale for each vessel segment, calcification, thrombolysis in myocardial infarction (TIMI) flow, collaterals, displaying the lesions and bifurcations.

OTHER OUTCOMES:
Safety Analysis | During coronary angiography
  The time(seconds), contrast usage(ml) and radiation dose(Gycm2) are recorded from the point of selective catheter engagement in the coronary ostium to the completion of the diagnostic study. The time, contrast and radiation to perform isocentering are included during dura-axis rotational coronary angiography. The time, contrast and radiation to engage the coronary ostium, exchange catheters, and perform non-coronary angiography are excluded from the analysis. All adverse events observed by the operator or reported by the patient are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Huiliang, M.D., Study Chair — General hospital of Chinese people's armed police forces; Jin Zhigeng, M.M., Study Director — General hospital of Chinese people's armed police forces; Yang Shengli, M.D., Principal Investigator — General hospital of Chinese people's armed police forces; Luo Jianping, M.M., Principal Investigator — General hospital of Chinese people's armed police forces; Ma Dongxing, M.D., Principal Investigator — General hospital of Chinese people's armed police forces; Liu Ying, M.M., Principal Investigator — General hospital of Chinese people's armed police forces; Han Wei, M.D., Principal Investigator — General hospital of Chinese people's armed police forces; Jing Limin, B.S.M., Principal Investigator — General hospital of Chinese people's armed police forces
Locations (1):
- General hospital of Chinese people's armed police forces, Beijing, China

REFERENCES:
- [Background] Garcia JA, Agostoni P, Green NE, Maddux JT, Chen SY, Messenger JC, Casserly IP, Hansgen A, Wink O, Movassaghi B, Groves BM, Van Den Heuvel P, Verheye S, Van Langenhove G, Vermeersch P, Van den Branden F, Yeghiazarians Y, Michaels AD, Carroll JD. Rotational vs. standard coronary angiography: an image content analysis. Catheter Cardiovasc Interv. 2009 May 1;73(6):753-61. doi: 10.1002/ccd.21918. PMID 19180661
- [Background] Klein AJ, Garcia JA, Hudson PA, Kim MS, Messenger JC, Casserly IP, Wink O, Hattler B, Tsai TT, Chen SY, Hansgen A, Carroll JD. Safety and efficacy of dual-axis rotational coronary angiography vs. standard coronary angiography. Catheter Cardiovasc Interv. 2011 May 1;77(6):820-7. doi: 10.1002/ccd.22804. Epub 2011 Mar 11. PMID 20853352
- [Background] Liu HL, Jin ZG, Yang SL, Luo JP, Ma DX, Liu Y, Han W. Randomized study on the safety and efficacy of dual-axis rotational versus standard coronary angiography in. Chin Med J (Engl). 2012 Mar;125(6):1016-22. PMID 22613524
- [Derived] Jin ZG, Bai R, Li Y, Yang Y, Han W, Zhao Q, Zhang L, Liu HL. Comparison of diagnostic accuracy of dual-axis rotational versus standard coronary angiography. Int J Cardiovasc Imaging. 2020 Feb;36(2):187-195. doi: 10.1007/s10554-019-01711-9. Epub 2019 Oct 18. PMID 31628576